CLINICAL TRIAL: NCT01572116
Title: Comparison the Effect of Lidocaine (With Epinephrine) With and Without Sufentanil on the Rate of Anesthesia of Intra-ligamentary Injection in Teeth With Irreversible Pulpitis
Brief Title: Effect of Sufentanil on the Rate of Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Mandana Abedi Tari, principal investigator, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRCT201110137790N1
Record Dates: First submitted 2012-03-03; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Irreversible Pulpitis
Keywords: sufentanil; irreversible pulpitis; intra ligament injection
MeSH Terms: interventions — Lidocaine; Epinephrine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine with Epinephrine+ Normal saline (Placebo Comparator)
  Interventions: Drug: Lidocaine with Epinephrine+ Normal saline
- Lidocaine with Epinephrine + sufentanil (Active Comparator)
  Interventions: Drug: Lidocaine with Epinephrine + sufentanil

INTERVENTIONS:
Drug: Lidocaine with Epinephrine+ Normal saline — PDL injection of 0/4 ml of lidocaine %2 with epinephrine,and Normal saline
  Arms: Lidocaine with Epinephrine+ Normal saline
Drug: Lidocaine with Epinephrine + sufentanil — PDL injection of 0/4 ml lidocaine with epinephrine and0/4 ml sufentanil ( 0/04 μg)
  Other Names: Brand name:Sufenta
  Arms: Lidocaine with Epinephrine + sufentanil

SUMMARY:
The aim of this study was to compare the effects of Lidocaine/epinephrine with and without Sufentanil on the rate of anesthesia after supplemental intraligamentary injection (PDL) in teeth with irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* patients in the age group of 18-65 years old
* healthy (ASA I, II)
* patients with first or second mandibular molars who need endodontic treatment
* vital tooth without a history of past endodontic treatment
* patients with clinical evidence of irreversible Pulpits with moderate to severe pain
* patients who signed consent form
* patients numbness at the lateral edge of the lips after inferior alveolar injection (INA) and those with positive respond to maximum output of pulp tester after INA.

Exclusion Criteria:

* pregnant or nursing
* necrotic tooth
* patients with allergy or contraindication toward non-opioid or opioid painkillers such as aspirin or NSAIDs
* Patients who have taken opioid or non opioid or steroid pain killers, antidepressants or sedative drugs in the past 48 hours
* patient with infectious diseases
* patient with moderate to sever periodontal disease
* those without numbness at the lateral edge of the lips after inferior alveolar injection (INA), and those do not respond to maximum output of pulp tester after INA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
depth of anesthesia | in different times such as :before the treatment,and during the treatment in these times: 1,5,9,13,17 minutes after starting the treatment
  The measuring method of the pain is Electric pulp tester

SECONDARY OUTCOMES:
intensity of the pain | before the treatment,Immediately after treatment, from commencement of treatment until complete pulpotomy stage, from commencement of treatment until initial file determination ,from commencement of treatment until end of pulpectomy
  The measuring method of the pain is Visual mentreatAnalogue Scale (VAS 0-170 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Abedi Tari, Dentist, Principal Investigator — Dental School of Azad University
Locations (1):
- Dental School of Azad University, Tehran, Tehran Province, Iran